CLINICAL TRIAL: NCT04349852
Title: Verbal Working Memory and Attention Remediation for Adults With Traumatic Brain Injury.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-00130
Record Dates: First submitted 2020-04-15; First posted 2020-04-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BrainHQ Cognitive Training Arm (Experimental): BrainHQ Cognitive Training Arm Participants will be randomized into the BrainHQ Cognitive Training modules which are 35 minute training sessions. There will be 30 training sessions. Since the intervention is presented both visually and verbally through the computer, and participants will be asked if they have a quiet space and noise cancelling headphones. Participants will complete the training protocols remotely and their performance will be tracked. Participants will complete the 30 training sessions remotely, but will meet with the study team member online prior to beginning the exercises and right after completing the session.
  Interventions: Behavioral: BrainHQ Cognitive Training Modules
- BrainHQ People Skills Arm (Other): Participants will be randomized into the BrainHQ's Brain Game exercises which are 35 minute training sessions. There will be 30 training sessions. Since the intervention is presented both visually and verbally through the computer, and participants will be asked to complete the training in a quiet space and time to complete these activities. Participants will complete the 30 training sessions remotely, but will meet with the study team member online each training session prior to beginning the exercises and right after completing the exercises.
  Interventions: Behavioral: BrainHQ People Skills Modules

INTERVENTIONS:
Behavioral: BrainHQ Cognitive Training Modules — The BrainHQ is a computerized training program developed from Posit Science designed to improve multiple cognitive domains. The subtests exercises include 6 modules for the experimental group: 1) Sound Sweeps: which is identify whether sound pitches are going up or down; 2) Memory Grids: matching pairs of words; 3) Syllable Stack: recognition of sequences of confusable syllables; 4) Fine Tuning: recognition of the order of confusable syllables; 5) To-Do List Training: reconstruction of sequences of verbal instructions; 6) In The Know: identification of details in a verbally presented story. Since the intervention is presented both visually and verbally through the computer, participants will be asked to complete their training in a quiet space and time to complete these activities.
  Arms: BrainHQ Cognitive Training Arm
Behavioral: BrainHQ People Skills Modules — The BrainHQ is a computerized training program developed from Posit Science designed to improve multiple cognitive domains. BrainHQ will provide 6 training modules for the control group: Crossword Puzzle - retrieve words according to the provided prompts. Lineup Four - Connect four colored discs so that they form a line in the horizontal, vertical or diagonal direction. Bricks Breaking Hex -Connect and remove bricks of the same color to clear the board. War Ship (Similar to Battleship)- place 5 vessels in the area at the left-hand side and sink enemy's hidden ships at the right-hand side by guessing enemy ship locations. Gem Swap - Form a line of 3 or more identical gems by swapping their positions. Sudoku - Fill each row, column, and 3x3 square with numbers 1 to 9 without repetition. Participants will spend 35 minutes at each training session. Participants will be asked to complete their training in a quiet space and time to complete these activities.
  Arms: BrainHQ People Skills Arm

SUMMARY:
This project will examine if computerized cognitive remediation will improve working memory and attention in 25 adults with a mild, moderate, or severe brain injury and compare their cognitive performance to the control group of 25 adults with a mild, moderate, or severe brain injury. The control group will train on computerized Brain Games. Participants in both groups will be assessed prior to training and immediately post-training and one month-post training.

DETAILED DESCRIPTION:
The study design will be randomized assignment with a control group. Participants in both groups will undergo three cognitive assessments at baseline, at the end of 30 cognitive training modules, and 1-month post-completion of the first follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Medically documented mild, moderate, or severe TBI;
* All subjects will be older than 18 years of age;
* Free from schizophrenia or bipolar disorder, due to the potential influence of such disorders on cognitive functioning;
* Free of current alcohol or drug abuse;
* At least 12 months post-injury.

Exclusion Criteria:

* Younger than 18 years old.
* A brain injury that is not medically documented.
* Being diagnosed with schizophrenia or bipolar disorder.
* Current alcohol or drug use diagnosis
* Less than 3 months post-injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in participants' logical memory after participating in BrainHQ training | baseline, 1 week post training, 4 weeks post training
  This will be measured by the Wechsler Memory Scale-IV (WMS-IV), Logical Memory subtest which is a measure of a person's ability to recall a story told to them.
Change in participants' verbal working memory after participating BrainHQ training | baseline, 1 week post training, 4 weeks post training
  This will be measured by the Auditory Consonant Trigram (ACT), the ACT is a standard assessment measure used to evaluate working memory, attention, and cognitive interference.
Change in participants' working memory after participating in BrainHQ training | baseline, 1 week post training, 4 weeks post training
  This will be measured by the Wechsler Memory Scale-IV (WMS-IV), Digit Span subtest which is a measure of working memory in which the person maintains their attention to the list of spoken numbers and ask to recall and state the list of numbers.
Participants' vocabulary after participating in BrainHQ training | baseline
  This will be measured by the Wechsler Adult Intelligence Scale IV, Vocabulary subtest which measure the ability to define specific words.
Participants' ability to recall information | baseline
  This will be measured by the Wechsler Adult Intelligence Scale IV, Information subtest which assesses the ability to recall general knowledge and acquired facts on different topics related to science, geography, and history.
Participants' abstract reasoning | baseline
  Measured by Wechsler Adult Intelligence Scale IV, Matrix Reasoning subtest which is a measure of abstract reasoning of visually presented stimuli.
Change in participants' level of reading | baseline, 1 week post training, 4 weeks post training
  This will be measured by Test of Premorbid Functioning which is a measure that reliably estimates levels of intelligence by asking the subject to read aloud the words on an established reading list.
Changes in the participants' processing speed | baseline, 1 week post training, 4 weeks post training
  This will be measured by Digit Symbol Modality Test which is a is a standard assessment measure used to measure processing speed, working memory, attention, and executive functioning. The standardized oral version will be administered.
Change in participants' verbal memory | baseline, 1 week post training, 4 weeks post training
  Measured by California Verbal Learning Test - II (CVLT). This test is a measure of verbal memory. A list of words is read aloud to the participants five times. After each list of words, the participant recalls the words. The participants will also be asked to recall the words from the list 20 minutes later.
Change in participants ability to assess auditory information | baseline, 1 week post training, 4 weeks post training
  This will be assessed with the Paced Auditory Serial Addition Test (PASAT) - 3 & 2 second versions which measures complex mental manipulation by adding the two most recent numbers that are presented auditorily. There are two sets of numbers that are presented at two different speeds. The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability.
Change in participants' verbal attention. | baseline, 1 week post training, 4 weeks post training
  Will be assessed with the Woodcock-Johnson - Understanding Directions subtest which is a measure of verbal attention. Participant are provided oral directions to point to different parts of pictures.
Change in participants' attention and verbal memory | baseline, 1 week post training, 4 weeks post training
  Actual Reality Performance test is a measure of attention and verbal memory, which requires the participants to follow directions and sequence steps of computerized task.
Changes to participants' ability to understand social cues | baseline, 1 week post training, 4 weeks post training
  Awareness of Social Inference Test (TASIT)- Short version: is a standard measure to recognize emotions and a speaker's intentions presented in a vignette.
Change in participants' sense of depression | baseline, 1 week post training, 4 weeks post training
  This will be self reported using the Beck's Depression Inventory - II. This is a standardized instrument for the assessment of depression with a self-report questionnaire.
Change in participants' sense of anxiety | baseline, 1 week post training, 4 weeks post training
  Measured by self reports with the Beck's Anxiety Inventory which is a self-report instrument for the assessment of anxiety.
Changes to participants' mental status | baseline, 1 week post training, 4 weeks post training
  Will be measured using the Lifetime Experience Questionnaire, \ a questionnaire to determine current and past mental.
Changes in participants' daily living | baseline, 1 week post training, 4 weeks post training
  The Functional Behavior Profile Questionnaire will be used to measure daily living status. This is a standardized questionnaire regarding activities of daily living, executive functioning, participation, problems solving and social relationships.
Changes in the pattern of participants social lifestyle | baseline, 1 week post training, 4 weeks post training
  This may be assessed with the Participation Assessment with Recombined Tools-Objective Questionnaire: A standardized questionnaire about social participation.
Changes in the participants' overall status | baseline, 1 week post training, 4 weeks post training
  Will be gauged by using the Promis Global Health Questionnaire. This is a standardized questionnaire that evaluates physical, mental and social health deficits common in people with brain injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Voelbel, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to gv23@nyu.edu. To gain access, data requestors will need to sign a data access agreement.